CLINICAL TRIAL: NCT07027319
Title: The Effect of Triple P Training Applied to Parents of Children With Autism Spectrum Disorder on Children's Repetitive Behaviors and Parents' Mood and Burnout Levels
Brief Title: The Effect of Triple P Training on Children's Repetitive Behaviors and Parents' Mood and Burnout Levels in Parents of Children With Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Özlem Teke (Other)
Collaborators: Uskudar University (Other)
Responsible Party: Sponsor-Investigator, Özlem Teke, MSc, Uskudar University
Organization: Uskudar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ozlem Teke
Record Dates: First submitted 2025-05-01; First posted 2025-06-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; positive parenting program; parent education; psychiatric nursing
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): This group will not be given any training other than the training they receive from the institution.
- Parenting Education (Experimental): The intervention group will receive 8 sessions of Triple P (positive parenting training).
  Interventions: Other: Parenting Education

INTERVENTIONS:
Other: Parenting Education — The intervention group will receive 8 sessions of Triple P (positive parenting training).
  Other Names: Triple P (Positive Parenting Program)
  Arms: Parenting Education

SUMMARY:
This project will be conducted in a private autism center in order to investigate the effects of Triple P training, which will be given to parents of children with Autism Spectrum Disorder, on the children's repetitive behaviors and the parents' burnout levels. The study is a randomized controlled trial and the study sample will consist of parents of children with Autism Spectrum Disorder. The children/parents included in the study sample will be numbered according to the order of arrival and 35 will be assigned to the intervention group and 35 will be assigned to the control group. During the randomization phase of the study, 70 children/parents with ASD will be randomly assigned to the intervention and control groups using Statistical Analysis Software. Data analysis will be performed using the Statistical Package for Social Sciences (SPSS v26.0, IBM Corp., Armonk, NY, USA). Descriptive data will be analyzed as mean, frequency and percentage. The conformity of quantitative data to normal distribution will be evaluated using the Kolmogorov-Smirnov test. Paired sample t-test will be used to compare dependent groups with normal distribution, independent sample t-test will be used to compare independent groups with normal distribution. P value will be considered significant if it is less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Having a child diagnosed with Autism Spectrum Disorder between the ages of 0 and 12
* Being willing to participate in the study
* Parents who speak Turkish

Exclusion Criteria:

* Parents of children with Autism Spectrum Disorder who are 13 years of age or older
* Parents who do not speak Turkish

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
General mental state of parents of children with autism spectrum disorder | T1: Baseline T2: 8 weeks T3: 3 months post-intervention
  General Health Questionnaire-28-Will be used to evaluate the general mental state of parents of children with autism spectrum disorder. The scale, developed by Goldberg and utilizing the "GSA-type scoring" method, is used as a four-item scale in which the first two items are scored negatively and the last two items positively. Accordingly, items a and b are scored as "0" (zero), while items c and d are scored as "1" (one). The total score on the scale can range from a minimum of 0 to a maximum of 28. Individuals who score 4 or below are considered to be "normal" in terms of mental health, whereas those who score 5 or above are evaluated as being in the "at-risk group" regarding their mental health.

OTHER OUTCOMES:
Assessment of repetitive behaviors in children with autism spectrum disorders | T1: Baseline T2: 8 weeks T3: 3 months post-intervention
  Repetitive Behavior Scale-Revised/RBS-R-It will be used to evaluate the repetitive behaviors of children with autism spectrum disorder and the severity of these behaviors. The items in the scale are rated using a four-point Likert scale (0: Behavior not present, 1: Mild level, 2: Moderate level, 3: Severe level). Higher scores on the scale are interpreted as indicating an increased severity of repetitive behaviors observed in children.
Burnout levels of parents of children with autism spectrum disorder | T1: Baseline T2: 8 weeks T3: 3 months post-intervention
  Parent Burnout Assessment (PBA)- Will be used to assess burnout levels of parents of children with autism spectrum disorder. The scale consists of 23 items and is scored using a 7-point Likert system. Higher total scores on the scale indicate greater severity of parental burnout. The possible score range for each item varies between 0 and 6.

CONTACTS AND LOCATIONS:
Overall Officials: Elçin Babaoğlu, Asst. Prof. Dr., Study Director — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share the pre-test, post-test and 3-month follow-up results obtained in the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: It is planned to be opened for access on 15.10.2025.
Access Criteria: It will be shared with researchers who contact the researcher.